CLINICAL TRIAL: NCT01703806
Title: Early Surgery Versus Conventional Treatment for Asymptomatic Patients With Severe Degenerative Mitral Regurgitation: A Propensity Analysis
Brief Title: Early Surgery Versus Conventional Treatment for Asymptomatic Severe Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Other Study IDs: 2007-0264
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Mitral Regurgitation
Keywords: Mitral regurgitation; Mitral valve repair; Watchful waiting
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Conventional Treatment: Patients in the conventional treatment group will be treated according to the 2006 ACC/AHA guidelines and they will be referred for surgery if they experience any symptoms, and referred for surgery if exertional dyspnea, LV ejection fraction <0.60, LV end-systolic dimension >40 mm, Doppler estimated pulmonary artery pressure > 50 mmHg, or atrial fibrillation develops.
  Interventions: Procedure: Watchful Observation
- Early Surgery: Patients in the early surgery group should undergo mitral valve surgery within 6 months of enrollment.
  Interventions: Procedure: Early Surgery

INTERVENTIONS:
Procedure: Early Surgery — MItral valve surgery
  Groups: Early Surgery
Procedure: Watchful Observation — Watchful observation
  Groups: Conventional Treatment

SUMMARY:
The timing of surgical intervention in asymptomatic patients with severe degenerative mitral regurgitation (MR) remains controversial. The benefit of early surgery has been suggested in prospective, observational studies, whereas a watchful waiting strategy seemed to be safe and effective in the other prospective study. The consensus guidelines for the performance of early surgery in asymptomatic patients with severe MR are different, reflecting controversy. Clinical outcome in asymptomatic patients with MR is poorly defined and it is important to identify high-risk patients in whom early surgery may be warranted. Thus, the investigators try to compare long-term outcomes of early surgery with those of a conventional-treatment strategy in a large prospective cohort of asymptomatic patients with severe degenerative MR using a propensity analysis, and to identify high-risk subgroups to whom early surgery is more beneficial.

DETAILED DESCRIPTION:
Surgery is the only definitive therapy for severe mitral regurgitation (MR) and the guidelines recommend surgery for management of MR to symptomatic patients or asymptomatic patients with left ventricular (LV) dysfunction. However, the timing of surgical intervention in asymptomatic patients with severe MR remains unclear due to the lack of randomized clinical trials comparing early surgery versus watchful waiting. The benefit of early surgery has been suggested in prospective, observational studies, whereas a watchful waiting strategy seemed to be safe and effective in the other prospective study. The consensus guidelines for the performance of early surgery in asymptomatic patients with severe MR are different, reflecting controversy. The 2006 American College of Cardiology/American Heart Association (ACC/AHA) guidelines recommend early surgery for asymptomatic patients if the success rate of mitral valve repair is expected to exceed 90%, but the 2007 European Society of Cardiology (ESC) guidelines recommend watchful waiting for such patients.

Clinical outcome in asymptomatic patients with MR is poorly defined and it is important to identify high-risk patients in whom early surgery may be warranted. Older patients and those with a larger effective regurgitant orifice (ERO) showed increased mortality under medical management, but it is controversial whether early surgery would improve clinical outcome of such patients, because the performance of surgery in high-risk patients might be associated with increased operative risk. Although randomized trials are required to establish indications for early surgery, ethical and financial constraints do not allow us to conduct a randomized trial and the investigators choose to perform a propensity analysis in a large prospective cohort of patients. The investigators try to compare long-term outcomes of early surgery with those of a conventional-treatment strategy that is based on current guidelines in a large prospective cohort of asymptomatic patients with severe degenerative MR using a propensity analysis, and examine the hypothesis that the reduction in cardiac mortality or cardiac event by early surgery is particularly evident among patients aged > 50 years or those with ERO ≥ 0.4 square centimeter.

All patients suspected of MR undergo transthoracic echocardiography. Entry evaluation includes demographic data, clinical presentation, physical findings and echocardiographic data. Eligibility is determined after a patient undergoes a thorough evaluation of clinical and echocardiographic data. After the eligible patient has signed informed consent, entry into the registry will take place. The treatment groups will not be randomly assigned and the choice of early surgery or conventional treatment for each patient is at the discretion of the attending physician, who explains the potential benefits of early surgery and procedural risks in detail and considers the preferences of individual patients most importantly. Patients in the early surgery group should undergo mitral valve surgery within 6 months of enrollment. Patients in the conventional treatment group will be treated according to the 2006 ACC/AHA guidelines and they will be educated to report immediately to a study coordinator or an investigator if they experience any symptoms, and referred for surgery if exertional dyspnea, LV ejection fraction <0.60, LV end-systolic dimension >40 mm, Doppler estimated pulmonary artery pressure > 50 mmHg, or atrial fibrillation develops. All patients will be followed at 3 months, 6 months, and 1 year; and at 6-month intervals thereafter until close-out of the study, and educated to call a study coordinator or an investigator if they experience any adverse events.

The Executive Committee will approve the final trial design and protocol. This committee will also be responsible for reviewing the final results, determining the methods of presentation and publication, and selection of secondary projects and publications. Members of the committee will include the PI and persons who will organize this study. The Data Safety Monitoring Board (DSMB) will review the safety data from this study and make recommendations based on safety analyses of serious adverse events and protocol deviation. The Clinical Events Committee will meet regularly to review and adjudicate all clinical events that occur throughout the study period. The statistical analysis will be performed according to the prespecified analysis plan as described in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic patients
* severe degenerative MR
* preserved left ventricular systolic function

Exclusion Criteria: According to the recommendations of the 2006 American College of Cardiology/American Heart Association (ACC/AHA) guidelines for surgical indications of severe MR, the criteria for exclusion from the study are defined as follows.

* patients with the presence of exertional dyspnea, or angina
* left ventricular ejection fraction < 0.60
* left ventricular end-systolic dimension > 40 mm
* atrial fibrillation
* significant aortic valve disease
* Doppler-estimated systolic pulmonary artery pressure > 50 mmHg
* patients who were not candidates for early surgery based on age > 80 years and coexisting malignancies
* patients who did not consent to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From1996 to 2016, 1000 consecutive, asymptomatic patients with severe degenerative MR who are potential candidates for early surgery, will be enrolled in the present study. Severe degenerative MR is defined as severe prolapse and/or flail leaflet of the mitral valve with an effective regurgitant orifice area > 0.40 square cm.
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Actual)
Dates: Start 1996-07 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2024-10 (Actual)

PRIMARY OUTCOMES:
Cardiac mortality | Up to 10 years
  Cardiac mortality is defined as operative mortality, sudden cardiac death, death from complications of myocardial infarction, heart failure, complications of cardiac intervention or other cardiac disease. Operative mortality is defined as death within 30 days of mitral valve surgery.

SECONDARY OUTCOMES:
Repeat mitral valve surgery | Up to 10 years
Hospitalization due to congestive heart failure | Up to 10 years
  A congestive heart failure hospitalization is defined as an unplanned, urgent admission for the management of congestive heart failure . A patient admitted for congestive heart failure have to show resting dyspnea and radiological signs of pulmonary edema and require intravenous diuretics.
A composite of cardiac events | Up to 10 years
  A composite of cardiac mortality, repeat MV surgery and hospitalization due to congestive heart failure during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Background] Kang DH, Kim JH, Rim JH, Kim MJ, Yun SC, Song JM, Song H, Choi KJ, Song JK, Lee JW. Comparison of early surgery versus conventional treatment in asymptomatic severe mitral regurgitation. Circulation. 2009 Feb 17;119(6):797-804. doi: 10.1161/CIRCULATIONAHA.108.802314. Epub 2009 Feb 2. PMID 19188506
- [Derived] Park SJ, Kim M, Son J, Jo HH, Kim GY, Kim J, Sun BJ, Kim EK, Lee S, Yoo JS, Yun SC, Jung SH, Song JM, Kang DH. Long-Term Outcomes of Early Surgery Versus Conventional Treatment for Asymptomatic Severe Mitral Regurgitation: A Propensity Analysis. Circulation. 2025 Oct 28;152(17):1209-1217. doi: 10.1161/CIRCULATIONAHA.125.074560. Epub 2025 Aug 13. PMID 40799133